CLINICAL TRIAL: NCT05204030
Title: Hashtag HPV: Engaging Parents Through Social Media to Increase HPV Vaccination
Brief Title: Hashtag HPV: HPV Vaccine Twitter Education Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Arkansas, Fayetteville (Other)
Collaborators: Thomas Jefferson University (Other); University at Albany (Other); National Cancer Institute (NCI) (NIH); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2108351667; 7R01CA229324-04 (NIH)
Record Dates: First submitted 2021-12-09; First posted 2022-01-24 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Human Papilloma Virus; Vaccine-Preventable Diseases
Keywords: Human Papilloma Virus; Human Papilloma Virus Vaccine; Human Papilloma Virus Vaccination; Intervention; Social media; Twitter; Parents; Child health; Cancer prevention; Vaccine acceptance; Narrative engagement; Patient self-report; Intention to vaccinate; community engagement; Public Health; Vaccination
MeSH Terms: conditions — Vaccine-Preventable Diseases

STUDY DESIGN:
Intervention Model Description: This 4-year study will evaluate the efficacy of a Twitter-based pilot intervention through a randomized controlled trial that will enroll a total of 600 parents/caregivers of children ages 9-14, whose child(ren) has not started the vaccine series. The intervention will consist of 2 arms and 12 monthly cohorts. After enrollment in the project, 300 participants will be randomized into the intervention arm and 300 participants will be enrolled into the control arm. Participants will be presented the intervention one month before their child's next wellcare visit.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrative (Experimental): The intervention condition will present narrative-focused messages about HPV and the HPV vaccine that includes important parent focused exemplar language and cultural norms on Twitter told through stories and characters (i.e., pseudo-parents).
  Interventions: Other: HPV Twitter Education Program - Narrative
- Non-Narrative (Active Comparator): The non-narrative condition will present scientific-focused messages about HPV and the HPV vaccine that includes important information relayed with numbers and facts.
  Interventions: Other: HPV Twitter Education Program - Non-Narrative

INTERVENTIONS:
Other: HPV Twitter Education Program - Narrative — This study will evaluate the efficacy of social media messages through Twitter, using a randomized controlled trial to determine what types of messages resonate with parents. The investigators will examine narrative messages (i.e., stories). The central hypothesis is that parents who read narrative-focused messages will be more likely to report narrative engagement, intention to vaccinate their child, and self-reported vaccination compared to parents who read non-narrative messages.
  Arms: Narrative
Other: HPV Twitter Education Program - Non-Narrative — This study will evaluate the efficacy of social media messages through Twitter, using a randomized controlled trial to determine what types of messages resonate with parents. The investigators will examine non-narrative messages (i.e., scientific information - numbers and facts). The central hypothesis is that parents who read narrative-focused messages will be more likely to report narrative engagement, intention to vaccinate their child, and self-reported vaccination compared to parents who read non-narrative messages.
  Arms: Non-Narrative

SUMMARY:
Parents use social media as an important parenting tool and source for health information. Using social media data to examine public opinion has had an early impact in public health and in cancer control and prevention efforts, including about the human papillomavirus (HPV) vaccine. A next step in this area of research is to develop and share messages on social media with parents to help inform and educate them about the HPV vaccine - ultimately assisting them with their decision to vaccinate their child. This study will evaluate the efficacy of social media messages through Twitter, using a randomized controlled trial to determine what types of messages resonate with parents. The investigators will examine differences between two types of messages - narrative messages (i.e., stories) and non-narrative messages (i.e., numbers and facts).

DETAILED DESCRIPTION:
Approximately 80 million people in the United States - or about one in four - are infected with human papillomavirus (HPV). HPV can cause cancer and there are vaccines that protect against cancer-related strains. Evidence supporting vaccine efficacy and safety is robust, and vaccine availability is widespread; however coverage rates continue to fall short of the national goal of 80% (48.6% in 2017). Understanding the barriers to vaccine acceptance, particularly related to parent resistance and their informational needs, is key to strengthening vaccine uptake among adolescents. Communicating evidence to parents and engaging them through narrative strategies may address some of the barriers during the decision-making process. Parents use social media as an important parenting tool and useful source for health information. In 2015, 75% of all parents used social media, and of these 1 in 4 used Twitter - equating to millions of parent users. The investigators know that using social media data for surveillance has had early impact in public health. However, what is not known is the effectiveness of using large-scale social media data to inform a targeted social media intervention to support HPV vaccine uptake. This study will advance the growing field by evaluating the efficacy of an innovative narrative-focused intervention designed to communicate evidence and information about the HPV vaccine for parents who use social media as a health information source. The approach is informed by narrative engagement theory that posits narratives strengthen knowledge and promote engagement through storytelling by tapping into feelings of empathy, identification, and transportation. The investigators will evaluate the efficacy of our Twitter-based pilot intervention in a randomized controlled trial that will enroll 600 parents/caregivers of children ages 9-14, whose child(ren) has not started the vaccine series. Our central hypothesis is that exposure to narrative-focused exemplar messages will lead to greater intention to vaccinate, and subsequently increased rates of vaccination in the intervention group compared to parents in the comparison group, who receive non-narrative HPV vaccine information (i.e., existing HPV vaccine information developed for Twitter). The investigators will use a Twitter-based Community Advisory Board, virtual focus groups, and existing Twitter messages developed by the HPV Roundtable to inform narrative-focused message development. The proposed study will address three specific aims: 1) Develop narrative-focused scientific exemplars for HPV vaccine communication utilizing existing online messages and community engagement on Twitter; 2) Quantify differences in engagement, intention to vaccinate, and self-reported vaccination between parents exposed to the narrative-focused scientific exemplars and parents exposed to non-narrative scientific messages; 3) Collect and analyze longitudinal participant metadata to measure Twitter activity during the study period. This study will impact the field of cancer prevention generally and HPV vaccination specifically by establishing the efficacy of narrative-focused health messaging campaign on social media, using a Twitter-based parent-engagement strategy.

ELIGIBILITY:
Inclusion Criteria: The study population includes parents who have children ages 9-14. All participants will be 18 years of age or older, and we will specifically target parents ages 25 and older. Eligibility for enrollment in the study will be limited to the following criteria:

1. Adults 18 years of age and older;
2. Utilizes Twitter, a social media platform;
3. Has a child aged 9-14;
4. Child has not started the 2-dose HPV vaccination series;
5. Has no child who has completed any dose HPV vaccination series;
6. Has a well-care visit scheduled for their child before December, 2022.

Exclusion Criteria:

1. Any adult who does not have a child 9-14 years of age;
2. Any adult who does not indicate some level of participation in Twitter;
3. Any adults who indicates a high level of anti-vaccine sentiment (assessed by vaccine hesitancy questions asked in the screener).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in caregiver self-reported HPV vaccination status of child questionnaire | Change in caregiver self-reported HPV vaccination of child at 1-month follow-up from baseline
  dependent variable; measure collects date of vaccination and number of vaccine doses to date
Change in caregiver self-reported HPV vaccination status of child questionnaire | Change in caregiver self-reported HPV vaccination of child at 1-year follow-up from 1-month follow-up
  dependent variable; measure collects date of vaccination and number of vaccine doses to date

SECONDARY OUTCOMES:
Caregiver self-reported empathy subscale adapted from Busselle & Bilandzic (2009) and Murphy, Frank, Chatterjee, Baezconde-Garbanati (2013). | only at 1-month post intervention
  mediating/moderating variable
Caregiver self-reported transportation subscale adapted from Murphy, Frank, Chatterjee, Baezconde-Garbanati (2013). Narrative versus Non-narrative: The Role of Identification, Transportation and Emotion in Reducing Health Disparities. | only at 1-month post intervention
  mediating/moderating variable
Caregiver self-reported identification subscale adapted from Murphy, Frank, Chatterjee, Baezconde-Garbanati (2013). Narrative versus Non-narrative: The Role of Identification, Transportation and Emotion in Reducing Health Disparities. | only at 1-month post intervention
  mediating/moderating variable
Change in caregiver self-reported intention to vaccinate their child questionnaire | Change in caregiver self-reported intention to vaccinate their child at 1-month follow-up from baseline
  dependent variable; measures readiness and likeliness to receive HPV vaccination
Change in caregiver self-reported intention to vaccinate their child questionnaire | Change in caregiver self-reported intention to vaccinate their child at 1-year follow-up from 1-month follow-up
  dependent variable; measures readiness and likeliness to receive HPV vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Massey, PhD, MPH, Study Director — University of California, Los Angeles
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Massey PM, Kearney MD, Hauer MK, Selvan P, Koku E, Leader AE. Dimensions of Misinformation About the HPV Vaccine on Instagram: Content and Network Analysis of Social Media Characteristics. J Med Internet Res. 2020 Dec 3;22(12):e21451. doi: 10.2196/21451. PMID 33270038
- [Background] Massey PM, Togo E, Chiang SC, Klassen AC, Rose M, Manganello JA, Leader AE. Identifying HPV vaccine narrative communication needs among parents on social media. Prev Med Rep. 2021 Jul 7;23:101488. doi: 10.1016/j.pmedr.2021.101488. eCollection 2021 Sep. PMID 34295614
- [Background] Massey PM, Chiang SC, Rose M, Murray RM, Rockett M, Togo E, Klassen AC, Manganello JA, Leader AE. Development of Personas to Communicate Narrative-Based Information About the HPV Vaccine on Twitter. Front Digit Health. 2021 Aug 4;3:682639. doi: 10.3389/fdgth.2021.682639. eCollection 2021. PMID 34713151